CLINICAL TRIAL: NCT03404804
Title: Oral Penicillin Challenge in the Pediatric Emergency Department
Brief Title: Oral Challenge in the Pediatric ED
Acronym: OPEN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, David Edward Vyles, Associate Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 1069530-3
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Penicillin Allergy; Pediatric Emergency Medicine
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral Challenge (Experimental): Patients with low-risk symptoms of amoxicillin allergy who receive oral amoxicillin to delabel their respective allergy.
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — Oral challenge with amoxicillin in patients who are deemed low-risk for true penicillin allergy

SUMMARY:
Our primary objective was to demonstrate the feasibility of utilizing a novel penicillin allergy questionnaire in the PED to identify a low-risk group of patients who will complete an oral challenge in the PED to test for an IgE-mediated allergic reaction. This was a 3-site pediatric emergency department study in which we challenged patients who met specific inclusion and exclusion criteria and were deemed low-risk.

Original aims included:

Aim 1: Demonstrate that a low-risk group of children with reported penicillin allergy will complete an oral penicillin challenge during a pediatric emergency department visit.

Aim 2: Conduct follow-up one day after oral challenge for all children and seven days after oral challenge for patients discharged with a prescription antibiotic to determine if a delayed or T-Cell mediated reaction occurs after exposure to multiple doses of penicillin or any other antibiotic prescribed at discharge.

Aim 3: Examine health care outcomes and prescription-related costs associated with illness treatment plans in children who are de-labeled as penicillin allergic after an oral challenge.

A secondary objective within the IRB protocol reports, "Our secondary objective is to examine whether health care outcomes and prescription-related costs are comparable between children who are de-labeled as penicillin allergic after an oral challenge compared to a standard of care group who are not challenged in the PED."

However, we never proceeded with enrolling patients with PCN allergy not challenged in the PED as it was planned for later in the study that did not come to fruition.

DETAILED DESCRIPTION:
A convenience sample of children aged 2 to 16 years who presented to the pediatric emergency department with a reported PCN allergy were administered an allergy questionnaire to determine risk-level designation. Low-risk eligible patients were offered an oral amoxicillin challenge. Differences among sites for family and provider interest in participation with oral challenges were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-16 with a parent/guardian (hereafter termed parent) reported history of allergy to a penicillin antibiotic in which the reported allergic reaction occurred at least six months prior to the current PED visit.
* Only children well enough to be discharged to home at the conclusion of the PED visit are eligible.

Exclusion Criteria:

* Children will be excluded if they have a history of developmental delay or inability to communicate the effects of an allergic reaction (non-verbal).
* Any contraindication to allergy testing will also result in exclusion
* (i.e. history of a severe allergic reaction to skin tests,,
* anaphylaxis in the past six weeks,
* known pregnancy
* child has a history of a condition that requires a beta blocker medicine for cardiac conditions, high blood pressure, migraine headaches, or eye drops for glaucoma (e.g. propranolol, metoprolol, atenolol and Timoptic®, or Betoptic® eye drops).
* Children who present to the PED with a rash, vomiting or current asthma symptoms including coughing, wheezing or breathing problems will also be excluded to ensure these do not mask reactions to an oral challenge.
* Patients deemed too acutely ill for participation (triage level 1 or 2 or as determined by the ED patient care team) will be excluded from the study.
* During this pilot study, we will exclude non-English speaking families. However, in subsequent studies we will include the non-English speaking population.
* Children who are wards of the state, in foster care or police custody or detention will be excluded.
* Children with any basal condition (trauma, infection, minor accidents, etc..) will be able to participate in the study provided they and their family are willing and do not meet the above-mentioned exclusion criteria.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2022-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David E Vyles, DO, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- David Vyles, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vyles D, Chiu A, Routes J, Castells M, Phillips EJ, Visotcky A, Fraser R, Pezzin L, Brousseau DC. Oral amoxicillin challenges in low-risk children during a pediatric emergency department visit. J Allergy Clin Immunol Pract. 2020 Mar;8(3):1126-1128.e1. doi: 10.1016/j.jaip.2019.09.022. Epub 2019 Oct 3. No abstract available. PMID 31586667

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible families were approached, consented, and then administered an allergy questionnaire. Research staff abstracted age and demographic characteristics from the medical record. Patients who met eligibility criteria and were deemed low-risk were offered an oral drug challenge with amoxicillin.
Pre-assignment Details: Here at CHW we documented 130 subjects who were only given the questionnaire to assess risk and were not oral challenged in the CHW ED. In March of 2020, the study questionnaire was adopted as standard of clinical care for any patients presenting with a history of penicillin allergy, thus the questionnaire portion of the study was no longer a research activity. However, if the assessed risk was low, patients were approached for participation in oral challenge and consented if agreeable
Groups:
- Oral Challenge: Patients getting amoxicillin
  Amoxicillin: Oral challenge with amoxicillin in patients who are deemed low-risk for true penicillin allergy
Period: Overall Study
Arm/Group | Oral Challenge
Started | 116 (116 participants consented and completed the oral amoxicillin challenge of this group.)
Completed | 116
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oral Challenge
Number analyzed (Participants) | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 116
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 67
  African American | 25
  Hispanic | 15
  unknown | 9
Region of Enrollment [Number; unit: participants]
  United States | 116

OUTCOME MEASURES:

1. Primary Outcome: Number of Oral Amoxicillin Challenge Participants Completing Challenge With Insignificant Adverse Result
Description: Demonstrate that a low-risk group of children with reported penicillin allergy will complete an oral penicillin challenge during a pediatric emergency department visit with insignificant adverse result.
Time Frame: 1 and 7 day followup phone surveys were conducted.
Population: Subjects who met inclusion/exclusion criteria, were confirmed to be low risk and agreed to be oral challenged.
Measure: Count of Participants; unit: Participants
Groups:
- Oral Challenge: Oral challenge with amoxicillin in patients who are deemed low-risk for true penicillin allergy
Arm/Group | Oral Challenge
Number analyzed (Participants) | 116
Participants
  Number of subjects who tolerated an oral challenge without demonstrating allergy. | 114
  Children who had mild symptoms after challenge deemed to be an allergic reaction. | 2

2. Secondary Outcome: Number of Participants With Oral Amoxicillin Challenge Follow-up to Determine if a Delayed or T-Cell Mediated Reaction Occurs After Exposure
Description: Conduct follow-up 6 months and 12 months after oral challenge for all children after oral challenge for patients discharged with a prescription antibiotic to determine if a delayed or T-Cell mediated reaction occurs after exposure to multiple doses of penicillin or any other antibiotic prescribed at discharge.
Time Frame: 6 months and 12 months after oral challenge
Population: Determined to be eligible by risk survey and giving consent to participate.
Measure: Count of Participants; unit: Participants
Groups:
- Oral Challenge: number of subjects who received an oral challenge.
Arm/Group | Oral Challenge
Number analyzed (Participants) | 116
Participants
  number of children who tolerated an oral amoxicillin challenge | 114
  Number of subjects who developed allergy symptoms. | 2

ADVERSE EVENTS:
Time Frame: 1 year after oral challenge.
Groups:
- Oral Challenge: Patients getting Oral challenge with amoxicillin in patients who are deemed low-risk for true penicillin allergy.
  Two children (1.7%) had mild symptoms after challenge deemed consistent with an allergic reaction by the PED provider. Four children experienced mild symptoms deemed not related to an allergic reaction by the examining physician
Arm/Group | Oral Challenge
All-Cause Mortality (participants affected / at risk) | 0/116
Serious Adverse Events (participants affected / at risk) | 0/116
Other Adverse Events (participants affected / at risk) | 2/116
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Challenge (N=116)
mild symptoms not related to allergic reaction to oral challenge (Skin and subcutaneous tissue disorders) | 2 (2) — Itching.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT03404804/Prot_SAP_001.pdf